CLINICAL TRIAL: NCT03477682
Title: Postoperative Management of Groin Flaps for Vascular Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-17005
Record Dates: First submitted 2018-03-05; First posted 2018-03-26 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Functional Status After Sartorius Flap of the Groin; Wound Complication
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The plastic surgeon who performs the sartorius flap does not know which group the patient will be randomized to (early ambulation versus standard 5 days bedrest) until after the surgery is completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Ambulation Group (Experimental): The patient will remain on bed rest for one day following surgery and will be encouraged to be out of bed and ambulating on the second day following surgery.
  Interventions: Other: Early ambulation
- Standard Group (No Intervention): The patient will remain on bed rest for five days following surgery and will be encouraged to be out of bed and ambulating on the sixth day following surgery.

INTERVENTIONS:
Other: Early ambulation — Patients who are in the experimental arm will have a shorter duration of bedrest restriction following sartorius surgery (1 day) versus the standard group (5 days bedrest).
  Arms: Early Ambulation Group

SUMMARY:
This is a randomized controlled trial designed to analyze the impact of bedrest duration on return to functional independence at discharge following sartorius flap for coverage of vascular reconstruction in the groin.

DETAILED DESCRIPTION:
This is a pilot prospective study with the purpose of evaluating the impact of bedrest duration on outcomes of groin muscle flaps used for groin coverage in patients undergoing open, infrainguinal vascular surgery. The investigators plan to target all patients undergoing groin muscle flaps for vascular groin coverage at UCSF.

All patients undergoing groin flaps will be block randomized into two cohorts: Cohort 1 - one day of bedrest (mobilize on post-op day 2) versus Cohort 2 - 5 days of bedrest (mobilize on post-op day 6).

The investigators perform approximately 50 infrainguinal muscle flaps per year. They aim to enroll 30 patients (15 per cohort).

Outcome measures include: surgical complication rates (including wound and lymphatic complications, readmissions, and reoperations), physical function, hospital length of stay, venous thromboembolism (VTE), and rates of discharge to a skilled nursing facility. The investigators will also examine the impact of bedrest on patient reported outcomes one month following surgery. Patient outcomes will be followed for 3 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing muscle flaps following infrainguinal, open vascular surgery. Patients must be ambulatory at baseline. Patients must be able to provide informed consent.

Exclusion Criteria:

* Patients who are unable to provide informed consent. Patients are non-ambulatory at baseline. Patients' clinical status is not amenable towards early ambulation. Enrollment is at the discretion of the vascular and plastic surgeons.
* Bilateral sartorius flaps

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in AM-PAC Score | 1 week
  AMPAC Score measures functional status

SECONDARY OUTCOMES:
Wound infection requiring medication | 3 months
  Described infection requiring antibiotics only, no surgery
Superficial wound dehiscence | 3 months
  Dehiscence of superficial layers (skin and subcutaneous tissue) requiring local wound care. Information will be gathered from medical record as charted by provider describing superficial wound dehiscence or via picture in the chart. This means separation at the skin level and may include, epidermis, dermis or subcutaneous fat or all three.
Deep wound dehiscence | 3 months
  Dehiscence of wound down to fascia, muscle, exposed vessels, requiring surgery. Information will be gathered from medical record as charted by provider or via picture. It will be described as wound dehiscence beyond the subcutaneous tissue down to fascia, muscle or exposed vessel and that required a re-operation by the plastic surgery team.
Wound infection requiring surgery | 3 months
  Wound infection or abscess requiring surgery (debridement, incision and drainage, exploration)
Length of hospital stay | 2 weeks
  Length of hospitalization following surgery, measured in days
Rehabilitation | 3 months
  Type of rehabilitation after surgery (home health, skilled nursing facility, home physical therapy, none)
SF36 Score | 3 months
  This survey measures quality of life and will be used to examine the impact of bedrest on patient reported quality of life outcomes postoperatively. Total scores range from 0-100 with higher scores indicating a more favorable state.
C-reactive protein | 1 week. Depending on the assigned group, this will be either on postoperative day two or six.
  A measure of nutritional status, measured on first day of mobilization
Albumin | 1 week. Depending on the assigned group, this will be either on postoperative day two or six.
  A measure of nutritional status, measured on first day of mobilization
Pre-albumin | 1 week. Depending on the assigned group, this will be either on postoperative day two or six.
  A measure of nutritional status, measured on first day of mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Hansen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenblatt DY, Rajamanickam V, Mell MW. Predictors of surgical site infection after open lower extremity revascularization. J Vasc Surg. 2011 Aug;54(2):433-9. doi: 10.1016/j.jvs.2011.01.034. Epub 2011 Mar 31. PMID 21458203
- [Background] Fischer JP, Nelson JA, Mirzabeigi MN, Wang GJ, Foley PJ 3rd, Wu LC, Woo EY, Kanchwala S. Prophylactic muscle flaps in vascular surgery. J Vasc Surg. 2012 Apr;55(4):1081-6. doi: 10.1016/j.jvs.2011.10.110. Epub 2011 Dec 29. PMID 22209610
- [Background] Genc A. Early mobilization of the critically ill patients: towards standardization. Crit Care Med. 2012 Apr;40(4):1346-7. doi: 10.1097/CCM.0b013e31823b8e44. No abstract available. PMID 22425834
- [Background] Fischer JP, Mirzabeigi MN, Sieber BA, Nelson JA, Wu LC, Kovach SJ, Low DW, Serletti JM, Kanchwala S. Outcome analysis of 244 consecutive flaps for managing complex groin wounds. J Plast Reconstr Aesthet Surg. 2013 Oct;66(10):1396-404. doi: 10.1016/j.bjps.2013.06.014. Epub 2013 Jul 5. PMID 23831123
- [Background] Evans GR, Francel TJ, Manson PN. Vascular prosthetic complications: success of salvage with muscle-flap reconstruction. Plast Reconstr Surg. 1993 Jun;91(7):1294-302. PMID 8497530
- [Background] Perme C, Chandrashekar R. Early mobility and walking program for patients in intensive care units: creating a standard of care. Am J Crit Care. 2009 May;18(3):212-21. doi: 10.4037/ajcc2009598. Epub 2009 Feb 20. PMID 19234100